CLINICAL TRIAL: NCT06549647
Title: Effect of Laser Acupuncture on Insulin Resistance in Obese Women With Polycystic Ovarian Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mena Faiez Shenouda, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005182
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo laser on acpoints + low caloric diet (Placebo Comparator): It will be consisted of 20 obese women diagnosed as having PCOS. Each will receive placebo laser on acupoints (3 sessions/week, 17 minutes/ session) in addition to low caloric diet for 3 months.
  Interventions: Other: low caloric diet; Other: Placebo laser acupoint stimulation
- Laser acupuncture + low caloric diet (Experimental): It will be consisted of 20 obese women diagnosed as having PCOS who will receive the same low caloric diet as in group (A) in addition to application of laser acupuncture on (REN 4,5), (ST 25,29,36,40), (CV 3,6,10,12),(SP 6), (L14), 1 minutes for each points (17 minutes/session), 3 times/week for 3 months.
  Interventions: Other: low caloric diet; Other: Laser Acupuncture

INTERVENTIONS:
Other: low caloric diet — A low caloric diet of 1200 Kcal will be followed by participant for 3 months. The dietary intervention follows a macronutrient ratio of 15% protein, 30% fat, and 55% carbohydrates. Participants are advised to consume 170-240g of complex carbohydrates, 60-100g of fat, and 55-93g of protein per day, with 20-35g of fiber. Patients are also advised to limit salt, tea, and caffeine intake, and receive supplemental vitamins to prevent deficiencies.
Other: Placebo laser acupoint stimulation — Placebo laser acupoint stimulation will be used for all participants in group (A).
  Arms: Placebo laser on acpoints + low caloric diet
Other: Laser Acupuncture — Eazyone EZ1 level laser will be used for the treatment procedures for all participants in group (B) only. Every participant in group (B) will be instructed briefly about the effect of laser acupoints therapy to gain her confidence and co-operation. It will be applied with infrared laser with 830 nm wavelength, 5 W power output and 0.5 J energy on the following acupoints while the patient lie in supine lying position. The head of the machine will be applied perpendicularly on each point for 1 min (17 min total), 3 times/ week for 4 weeks.
  Arms: Laser acupuncture + low caloric diet

SUMMARY:
This study will be conducted to investigate the effect of laser acupuncture on insulin resistance in obese women with polycystic ovarian syndrome.

DETAILED DESCRIPTION:
Women with Polycystic Ovary Syndrome (PCOS) face an increased risk of various health issues, including glucose intolerance, type 2 diabetes, hypertension, dyslipidemia, and subfertility. The prevalence of insulin resistance (IR) in PCOS can range from 44% to 70%, with longitudinal studies indicating that worsening IR over time in obese women with PCOS is associated with an increased risk of early-onset type 2 diabetes.

Conventional interventions, such as oral contraceptives, metformin, and hormonal therapy, have been developed to address the effects of PCOS. However, these treatments can have adverse side effects, including an increased risk of estrogen-related cancers. Consequently, lifestyle modifications to prevent aberrant immune activation and minimize exposure to inflammatory agents have emerged as a more sustainable approach.

Emerging evidence suggests the potential of alternative physical therapy modalities, such as transcutaneous electrical nerve stimulation, electro-acupuncture, and laser acupuncture, in managing PCOS. Laser acupuncture, in particular, has been shown to reduce sympathetic activity, decrease ovarian androgen release, and modulate the activity of higher centers, ultimately influencing gonadotropin-releasing hormone secretion and the menstrual cycle. Additionally, laser acupuncture may reduce the levels of pro-inflammatory cytokines, which contribute to insulin resistance and atherosclerosis.

While a few studies have investigated the effects of laser acupuncture on insulin resistance in obese women with PCOS, further research is needed to provide deeper insights into the benefits of this intervention and its role in managing insulin resistance in this population, which could expand the clinical applications of laser therapy in physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Forty obese women with PCOS as clinically diagnosed by gynecologist.
* Their ages will be ranged from 20 to 35 years old.
* Their BMI will be ranged from 30-40 kg/m2
* Their waist/hip ratio will be >0.8
* All of them should have at least two criteria of the Rotterdam diagnostic criteria of PCOS.

Exclusion Criteria:

* Cushing syndrome, diabetes mellitus, Thyroid dysfunction, Hypothalamic amenorrhea, Ovarian hyperplasia
* Respiratory, renal and liver dysfunction.
* Skin diseases and any other condition that may prevent the usage of laser (skin cancer, active acne and skin infections).
* Malignancy

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Body mass index (BMI) | 3 months
  It will be calculated from the weight and height of each participant in both groups (A&B), before beginning of the study and after end of the study program, according to the following equation:
  BMI =(Weight (kg))/(Height square (m²)) kg/m²
Waist/hip ratio | 3 months
  It will be calculated from the waist and hip circumferences for all participants in both groups (A&B) according to the equation waist/hip ratio= (waist / hip) before and after the end of study.
Oral glucose tolerance test | 3 months
  A venous blood sample will be collected from each participant before and after the end of study. The 2-hour plasma glucose level <140 mg/DL (7.8 MMOL/L) is considered normal. A blood glucose level between 140 and 199 mg/DL (7.8 and 11 MMOL/L) is considered impaired glucose tolerance, or pre-diabetes.
Fasting plasma insulin | 3 months
  A venous blood sample will be collected from each participant before and after the end of study. Fasting plasma insulin level will be measured for all participants in both groups (A&B) after at least 8 hours of fasting. Normal insulin level is 3-8µIU/ml, mild insulin resistance is 8-10µIU/ml, moderate insulin resistance is 10-12µIU/ml and sever insulin resistance is >12 µIU/ml.
Glucose /insulin ratio | 3 months
  A venous blood sample will be collected from each participant before and after the end of study. A G/I ratio of less than 4.5 has been shown to be sensitive and specific for insulin resistance in a group of women with PCOS.
Homeostasis Model Assessment (HOMA IR) | 3 months
  It will be calculated for all participants in both groups (A&B) before and after the end of the treatment according to the following equation: HOMA-IR = insulin (MU/L) × glucose (mmol/L)/22.5. HOMA-IR ≥2.5 should be considered a reasonable indicator of insulin resistance.

SECONDARY OUTCOMES:
Polycystic Ovary Syndrome Quality of Life scale (PCOSQ) | 3 months
  The quality of life of participants in both groups (A & B) will be assessed before and after the treatment program using a 26-item questionnaire divided into five sections: emotions (8 items), body hair (5 items), weight concerns (5 items), infertility concerns (4 items), and menstrual irregularities (4 items). Each item is rated on a seven-point scale, where 7 indicates the best situation and 1 the worst. Scores are calculated as means for each domain, with total scores categorized into four intervals reflecting varying effects on quality of life.Ultimately, the first interval values (from 1 to < 3 points) represent marked effects on quality of life; second interval values (from 3 to < 4 points) represent the marginal effect on quality of life; third interval values (from 4 to < 5 points) represent the minimal effect on quality of life; fourth interval (5 points) represents no effect on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Azza Barmoud Nashed Kassab, PhD, Study Chair — Professor of Physical Therapy for Woman's Health, Cairo University